CLINICAL TRIAL: NCT02013856
Title: The Effects of Apple Derived Flavanols on Cardiovascular Disease Risk
Brief Title: The Effects of Apple Derived Flavanols on Cardiovascular Disease Risk (FLAVASCULAR Study)
Acronym: FLAVASCULAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Quadram Institute Bioscience (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: IFR05/2013
Record Dates: First submitted 2013-12-09; First posted 2013-12-17 (Estimated); Last update posted 2016-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Blood Pressure
Keywords: Blood pressure; Flavanols; Cardiovascular disease
MeSH Terms: conditions — Cardiovascular Diseases | interventions — procyanidin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Low Epicatechin and procyanidin (Experimental): Low epicatechin and procyanidin doses
  Interventions: Dietary Supplement: Low Epicatechin and procyanidin
- High Epicatechin and procyanidin (Experimental): High epicatechin and procyanidin doses
  Interventions: Dietary Supplement: High Epicatechin and procyanidin
- High Procyanidin (Experimental): High procyanidin only
  Interventions: Dietary Supplement: High procyanidin
- Placebo (Placebo Comparator): No epicatechin and procyanidin
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Low Epicatechin and procyanidin — 70 mg epicatechin and 65 mg procyanidins once daily for 28 days
  Arms: Low Epicatechin and procyanidin
Dietary Supplement: High Epicatechin and procyanidin — 140 mg epicatechin and 130 mg procyanidins once daily for 28 days
  Arms: High Epicatechin and procyanidin
Dietary Supplement: High procyanidin — No epicatechin and 130 mg procyanidins once daily for 28 days
  Arms: High Procyanidin
Dietary Supplement: Placebo — Placebo control once daily for 28 days
  Arms: Placebo

SUMMARY:
Fruit and vegetable rich diets are associated with a reduced risk of cardiovascular disease (CVD). The protective effect may be ascribed to compounds contained within these foods, called flavonoids. Flavanols (epicatechin and procyanidins) are a particular group of flavonoids and are found mostly in apples, berry fruits, dark chocolate, tea and red wine. There is evidence to suggest that ingestion of flavanol rich foods and beverages beneficially alter 'markers' of CVD risk (e.g. blood pressure). The aim of this study is to determine the acute and chronic effects of apple derived flavanols on some risk markers for CVD.

DETAILED DESCRIPTION:
This study is a single arm randomized, 4-phase crossover design.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ≥ 50 years of age
* Systolic blood pressure 130 - 159 mmHg

Exclusion Criteria:

* History of cardiovascular events such as stroke, myocardial infarction trans- ischaemic attacks or peripheral vascular disease
* Kidney or liver disease/problems
* Diabetes
* Asthmatics (unless no medication taken for 1 year - occasional use will be assessed on an individual basis)
* Prescribed anti-hypertensive medication
* HRT (unless the participant has used the therapy for ≥ 6 months)
* Lipid lowering therapies e.g. statins
* Other medications that may affect any of the study outcome measures e.g. vasodilators (this will be assessed on a case by case basis)
* Current smoker (or stopped for less than 3 months)
* Throat surgery or neck injury
* Allergy to apples
* Consumption of fish oil supplements unless willing to discontinue them up for 4 weeks preceding the start of the study and for the duration of the study. (All other supplements will be assessed on a case by case basis)
* Gastro-intestinal diseases (excluding hiatus hernia unless symptomatic or study intervention/procedure is contra-indicated).
* Parallel participation in another research project which involves dietary intervention
* Participation in another research project which has involved blood sampling within the last four months unless the total amount of combined blood from both studies does not exceed 470 ml.
* Has donated or intends to donate blood within 16 weeks prior to or during the study period.
* Depressed or elevated blood pressure measurements (<90/50 or 95/55 if symptomatic or >160/100 (mmHg)) during the course of the trial.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2014-07; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Changes in systolic blood pressure from baseline | Baseline, 2 hours and 4 weeks

SECONDARY OUTCOMES:
Changes in plasma lipid profile from baseline | Baseline and 4 weeks
Change in plasma endothelin-1 from baseline | Baseline and 4 weeks
Changes in plasma nitric oxide metabolites from baseline | Baseline, 2 hours and 4 weeks
Changes in blood glucose from baseline | Baseline and 4 weeks
Changes in pulse wave velocity from baseline | Baseline, 2 hours and 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Paul Dr Kroon, PhD, Principal Investigator — Quadram Institute Bioscience
Locations (1):
- Institute of Food Research, Norwich, Norfolk, United Kingdom

REFERENCES:
- [Derived] Hollands WJ, Tapp H, Defernez M, Perez Moral N, Winterbone MS, Philo M, Lucey AJ, Kiely ME, Kroon PA. Lack of acute or chronic effects of epicatechin-rich and procyanidin-rich apple extracts on blood pressure and cardiometabolic biomarkers in adults with moderately elevated blood pressure: a randomized, placebo-controlled crossover trial. Am J Clin Nutr. 2018 Nov 1;108(5):1006-1014. doi: 10.1093/ajcn/nqy139. PMID 30475960